CLINICAL TRIAL: NCT01640574
Title: Randomised Parallel Open Label Comparison Between 7 and 14 Day Primaquine Combined With 3-day Dihydroartemisinin-piperaquine or 3-day Chloroquine Regimens for Radical Cure of Plasmodium Vivax
Brief Title: Comparison Between 7 and 14 Day Primaquine Combined With Dihydroartemisinin-piperaquine or 3 Day Chloroquine Radical Cure of P. Vivax (BPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMRU1102
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Vivax Malaria
Keywords: Vivax; Chloroquine; Primaquine; Dihydroartemisinin-Piperaquine
MeSH Terms: conditions — Malaria, Vivax | interventions — Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- DHA-P 7 days (Experimental): Dihydroartemisinin-piperaquine + Primaquine: DHA-P 7mg/kg/day dihydroartemisinin and 55mg/kg/day piperaquine daily for 3 days and Primaquine 1 mg/kg once daily for 7 days
  Interventions: Drug: Dihydroartemisinin-Piperaquine
- DHA-P 14 days (Experimental): Dihydroartemisinin-piperaquine + Primaquine: DHA-P 7mg/kg/day dihydroartemisinin and 55mg/kg/day piperaquine daily for 3 days Primaquine 0.5 mg/kg daily for 14 days
  Interventions: Drug: Dihydroartemisinin-Piperaquine
- Chloroquine 7 days (Active Comparator): Chloroquine + Primaquine: Chloroquine 10, 10, 5 and Primaquine 1 mg/kg once daily for 7 days
  Interventions: Drug: Chloroquine
- Chloroquine 14 days (Active Comparator): Chloroquine + Primaquine: Chloroquine 10, 10, 5 and Primaquine 0.5 mg/kg daily for 14 days
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Dihydroartemisinin-Piperaquine — Dihydroartemisinin-piperaquine + Primaquine: DHA-P 7mg/kg/day dihydroartemisinin and 55mg/kg/day piperaquine daily for 3 days and Primaquine 1 mg/kg once daily for 7 days
  Arms: DHA-P 7 days
Drug: Dihydroartemisinin-Piperaquine — Dihydroartemisinin-piperaquine + Primaquine: DHA-P 7mg/kg/day dihydroartemisinin and 55mg/kg/day piperaquine daily for 3 days Primaquine 0.5 mg/kg daily for 14 days
  Arms: DHA-P 14 days
Drug: Chloroquine — Chloroquine + Primaquine: Chloroquine 10, 10, 5 and Primaquine 1 mg/kg once daily for 7 days
  Arms: Chloroquine 7 days
Drug: Chloroquine — o Chloroquine + Primaquine: Chloroquine 10, 10, 5 and Primaquine 0.5 mg/kg daily for 14 days
  Arms: Chloroquine 14 days

SUMMARY:
In Southeast Asia, Plasmodium vivax (Pv) infection reaches 50-80% and bears a greater burden of disease than Plasmodium falciparum (Pf). As control over Pf improves, Pv will assume increasingly larger percentages of malaria prevalence. The chronicity of Pv, due to the latent liver stage (hypnozoite) not eradicated by chloroquine, causes recurring disability and compounds the economic burden of those with symptomatic disease. The only widely available treatment for hypnozoites is primaquine, which, because of challenges with tolerability, safety in G6PD deficient persons, and compliance, is not commonly prescribed for the treatment of Pv. Currently, chloroquine is used for the treatment of the blood stages of Pv, however, there are concerns about increasing parasite resistance. Alternative treatments, such as artesunate, should be considered in the future of the treatment of blood stage Pv. The use of primaquine in the treatment of hypnozoites (radical cure) should be emphasized so that transmission of Pv can be controlled.

This study aims to determine the optimal primaquine regimen for radical cure of Plasmodium vivax. Chloroquine is currently the standard of treatment for Plasmodium vivax. Chloroquine may have synergistic effects when used with primaquine and due to its long half-life may delay the first relapse of vivax malaria. In contrast, artesunate does not have documented interactions with primaquine and has a very short half-life, thus, presumably will have no impact on first relapse. Combining primaquine with these two anti-malarials may lead to an alternative regimen for Pv infection and changing the primaquine dosing regimen may lead to a more practical and efficacious therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 months old
* Microscopic diagnosis of Plasmodium vivax malaria mono-infection
* Participant or parent/guardian is willing and able to give informed consent for participation in the study
* Able (in the Investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Severe malaria
* History of allergy or adverse reaction to artesunate, piperaquine, chloroquine, or primaquine
* Blood transfusion in the past 3 months
* G6PD deficiency by rapid test
* Hematocrit ≤ 25%
* Pregnancy at the time of screening
* Breastfeeding an infant < 6 months old
* Presence of any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2012-02; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Recurrence of P. vivax | 52 weeks
  Recurrence with Plasmodium vivax malaria within 52 weeks of first treatment dose

SECONDARY OUTCOMES:
Adverse Events | 28 days
  Number of adverse events within 28 days of study medication
Recurrence of P. vivax | 6 months
  Recurrence with Plasmodium vivax malaria within 6 months of first treatment dose
Drug concentrations | 63 days
  Chloroquine, piperaquine and primaquine drug levels

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, MD, Principal Investigator — University of Oxford; Cindy Chu, MD, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

REFERENCES:
- [Derived] Stadler E, Cromer D, Mehra S, Adekunle AI, Flegg JA, Anstey NM, Watson JA, Chu CS, Mueller I, Robinson LJ, Schlub TE, Davenport MP, Khoury DS. Population heterogeneity in Plasmodium vivax relapse risk. PLoS Negl Trop Dis. 2022 Dec 19;16(12):e0010990. doi: 10.1371/journal.pntd.0010990. eCollection 2022 Dec. PMID 36534705
- [Derived] Chu CS, Watson JA, Phyo AP, Win HH, Yotyingaphiram W, Thinraow S, Soe NL, Aung AA, Wilaisrisak P, Kraft K, Imwong M, Hanpithakpong W, Blessborn D, Tarning J, Proux S, Ling C, Nosten FH, White NJ. Determinants of Primaquine and Carboxyprimaquine Exposures in Children and Adults with Plasmodium vivax Malaria. Antimicrob Agents Chemother. 2021 Oct 18;65(11):e0130221. doi: 10.1128/AAC.01302-21. Epub 2021 Aug 16. PMID 34398667
- [Derived] Chu CS, Phyo AP, Turner C, Win HH, Poe NP, Yotyingaphiram W, Thinraow S, Wilairisak P, Raksapraidee R, Carrara VI, Paw MK, Wiladphaingern J, Proux S, Bancone G, Sriprawat K, Lee SJ, Jeeyapant A, Watson J, Tarning J, Imwong M, Nosten F, White NJ. Chloroquine Versus Dihydroartemisinin-Piperaquine With Standard High-dose Primaquine Given Either for 7 Days or 14 Days in Plasmodium vivax Malaria. Clin Infect Dis. 2019 Apr 8;68(8):1311-1319. doi: 10.1093/cid/ciy735. PMID 30952158
- [Derived] Chu CS, Bancone G, Moore KA, Win HH, Thitipanawan N, Po C, Chowwiwat N, Raksapraidee R, Wilairisak P, Phyo AP, Keereecharoen L, Proux S, Charunwatthana P, Nosten F, White NJ. Haemolysis in G6PD Heterozygous Females Treated with Primaquine for Plasmodium vivax Malaria: A Nested Cohort in a Trial of Radical Curative Regimens. PLoS Med. 2017 Feb 7;14(2):e1002224. doi: 10.1371/journal.pmed.1002224. eCollection 2017 Feb. PMID 28170391